CLINICAL TRIAL: NCT07072078
Title: The Effect of Video-Based Communication on Reducing Loneliness in Intensive Care Unit Patients: A Quasi-Experimental Study
Brief Title: The Role of Nurses in Video-Based Communication to Reduce Loneliness in Intensive Care Unit Patients
Acronym: VBC-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NURS-202506.01
Record Dates: First submitted 2025-06-29; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Loneliness During COVID-19; Loneliness
Keywords: Loneliness; Intensive Care Unit; Video-based Communication

STUDY DESIGN:
Intervention Model Description: This study used a parallel design with two groups: an intervention group and a control group. A total of 36 ICU patients were randomly assigned to each group (18 participants per group). The intervention group received video-based communication with family members once daily for three consecutive days, with each session lasting 5 to 20 minutes. The control group received standard ICU care without the intervention. Loneliness was measured in both groups using the De Jong Gierveld Loneliness Scale before and after the intervention. The study aimed to assess the effectiveness of video-based communication in reducing emotional and social loneliness among ICU patients.
Masking Description: This was an open-label study. No parties were masked. All participants, care providers, and investigators were aware of the group assignments and interventions being administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - Video-based Communication (Experimental): Participants in this group received structured video-based communication with their family members using WhatsApp. Each session lasted 5-20 minutes and was conducted once daily for three consecutive days. The communication was facilitated by a nurse and included positive messages, emotional support, and discussion of future plans. The aim was to reduce emotional and social loneliness in ICU patients.
  Interventions: Behavioral: Video-based Communication
- Control Group - Standard ICU Care (No Intervention): Participants in this group received standard ICU care without any video-based communication intervention. They continued with routine treatment and monitoring in the ICU setting for the duration of the study period. This group was used as a comparison to assess the impact of video-based communication on loneliness levels.

INTERVENTIONS:
Behavioral: Video-based Communication — Participants received structured video-based communication sessions with their family members using the WhatsApp platform. The intervention was delivered once daily for three consecutive days, with each session lasting between 5 and 20 minutes. Communication was guided to include emotional support, positive conversations, and future-oriented discussion. The sessions were facilitated by nurses who ensured clinical stability, technical setup, and emotional readiness of the patient. This intervention aimed to reduce emotional and social loneliness among ICU patients and was integrated into standard intensive care routines without disrupting medical care.
  Arms: Intervention Group - Video-based Communication

SUMMARY:
This study aims to evaluate the effectiveness of video-based communication in reducing loneliness among intensive care unit (ICU) patients at Dr. Hasan Sadikin General Hospital in Bandung, Indonesia. ICU patients often experience psychological distress, particularly loneliness, due to restricted family visits and physical isolation.

A quasi-experimental design with a pre-test and post-test control group is used, involving 36 participants who are randomly assigned to either the intervention or control group. The intervention group receives structured video-based communication with family members for three consecutive days, with each session lasting between 5 to 20 minutes. Nurses facilitate the intervention by ensuring patient safety, providing emotional support, and assisting with the communication process. The control group receives standard ICU care without the communication intervention.

Loneliness levels are assessed using the De Jong Gierveld Loneliness Scale (DJGLS) before and after the intervention.

DETAILED DESCRIPTION:
This study investigates the effectiveness of video-based communication in reducing loneliness among patients in the Intensive Care Unit (ICU). Loneliness is a common psychosocial issue in ICU patients, caused by physical isolation, limited visitation policies, and minimal social interaction. It is associated with increased stress, potential suppression of immune response, and extended hospitalization. The intervention provides a practical approach by enabling virtual interaction with family members, allowing emotional connection despite physical distance.

The study uses a quasi-experimental design with a pre-test and post-test control group. A total of 36 patients are recruited from Dr. Hasan Sadikin General Hospital in Bandung and randomly assigned to either an intervention or control group. The intervention group receives structured video-based communication using WhatsApp for three consecutive days, with each session lasting between 5 and 20 minutes. The control group receives standard ICU care without the additional communication support. The De Jong Gierveld Loneliness Scale (DJGLS) is used to assess emotional and social loneliness levels before and after the intervention.

Nurses act as primary facilitators in the intervention. Their responsibilities include ensuring clinical stability, setting up the communication devices, emotionally supporting patients during the sessions, monitoring patient responses, documenting the process, and coordinating communication with family members.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to the intensive care unit (ICU)
2. Patients aged over 18 years with a minimum of 72 hours of care in the ICU
3. Patients who are able to understand and communicate in the Indonesian language

Exclusion Criteria:

1. Patients with medical conditions such as decreased consciousness, total blindness, or severe neurological disorders
2. Patients with a history of psychiatric disorders

Drop Out:

1. Patients who are discharged from the ICU of Dr. Hasan Sadikin General Hospital during the study period will be considered drop-outs
2. Patients whose health deteriorates to the extent that they are unable to continue participation in the study
3. Patients who die during the study period
4. Patients who are transferred from the ICU to general inpatient wards

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-12-24 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Change in Loneliness Score (De Jong Gierveld Loneliness Scale) | Baseline (Day 1) to Post-Intervention (Day 3)
  This outcome measures the change in loneliness among ICU patients before and after the intervention, using the De Jong Gierveld Loneliness Scale (DJGLS). The scale assesses both emotional and social loneliness with 11 items, validated in Indonesian. Higher scores indicate greater loneliness. The score is recorded at baseline (pre-intervention) and after 3 days of intervention (post-test). The difference in mean scores is used to assess effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Cecep Eli Kosasih, S.Kp., MNS., Ph.D, Principal Investigator — Universitas Padjadjaran; Ristina Mirwanti, S.Kep., Ners., M.Kep., Study Director — Universitas Padjadjaran
Locations (1):
- dr. Hasan Sadikin General Hospital, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No